CLINICAL TRIAL: NCT06602908
Title: Functional Status for Surgically and Non-surgically Treated Patients With Acute Achilles Tendon Rupture Following a Public Municipal Rehabilitation - A Prospective Cohort Study
Brief Title: Functional Status for Surgically and Non-surgically Treated Patients With Acute Achilles Tendon Rupture Following a Public Municipal Rehabilitation
Status: Active, not recruiting | Type: Observational
Sponsor: Københavns Kommune (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jonas Samsø Larsen, Principal investigator. Cand. scient phys. University of Southern Denmark. Developmental physiotherapist, Centre of Rehabilitation Copenhagen City, Denmark, University of Southern Denmark
Other Study IDs: F-24036357
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-04

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles Tendon Rupture; Cohort Study; Functional Status; Heel Rise Tests; Associating Factors; Public Municipal Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surgically and non-surgically treated patients with achilles tendon rupture: One hundred patients with surgically and non-surgically treated achilles tendon rupture referred to rehabilitation in the municipality of Copenhagen.

SUMMARY:
A total Achilles tendon rupture is a common injury most often occuring in people aged between 30 and 50 years. The injury is more common amongst men than women (ratio 3:1) and typically occur during sports activities involving excentric and/or plyometric muscle work in plantar flexion of the foot (e.g., jumping, sprinting, change of directions).

Overall, there is no significant difference in treatment outcomes between surgical and non-surgical treatment besides a slightly greater risk of adverse events in surgical treatment and a small increased risk of re-rupture in non-surgical treatment. Several studies have investigated the importance of rehabilitation protocols without outcome differences between groups comparing more or less aggressive strategies.

Achilles tendon rupture often leads to significant limitations in functional level. Some of the most common used outcome measures for functional status are the heel rise tests evaluating endurance and maximum heel rise height. Studies using these tests often shows substantial deficits several years after the injury.

The purpose of this study is to investigate factors associated with functional status after rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient has an acute achilles tendon rupture (treated within 14 days after injury).
* Adult patients aged of 18 years or older.
* Patients has given informed consent to participate in the study.

Exclusion Criteria:

* Patients with bilateral achilles tendon rupture
* Patients with re-rupture of previous achilles tendon rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgically and non-surgically treated achilles tendon rupture referred to rehabilitation in the municipality of Copenhagen.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional test battery: Heel rise test for endurance and maximal height | LSI is measured at the final visit during rehabilitation (Often 6 months from injury or operation). Further assessment 12 months follow up from injury or operation.
  Heel rise test for endurance:
  One legged heel rise test performed in standing position barefooted on the floor with fingertips placed against the wall for balance.
  Number of repetitions until failure is counted on non-injured leg and afterwards on injured leg. The difference between injured leg and non-injured leg is measured by
  Limb Symmetry Index in % (LSI):
  (injured leg)/(non-injured leg) x 100
  Heel rise test for maximal height:
  One legged heel rise test performed in standing position barefooted on the floor with fingertips placed against the wall for balance.
  The patient is instructed to go as high as possible. The height from the floor until the distal end of calcaneus is measured with a tape measure to the nearest 0.1 cm.
  The difference between injured leg and healthy leg is measured by
  Limb Symmetry Index in % (LSI):
  (injured leg)/(non-injured leg) x 100

SECONDARY OUTCOMES:
Patient Specific Functional Score (PSFS) | Change from baseline to the final visit of rehabilitation (Often 6 months from injury or operation). Further assessment 12 months follow up from injury or operation.
  Patients are asked to identify 5 activities they are having difficulty with as a result of their current problem.
  Each activity is scored on a 0 (unable to perform activity) to 10 (able to perform activity at same level as before injury or problem) points numeric rating scale.
  An average Patient-Specific Functional Scale (PSFS) score is calculated and can vary from 0 to 10, with higher scores representing higher levels of lower extremity functional status.
Pain Numeric Rating Scale (NRS) | Change from baseline to the final visit of rehabilitation (Often 6 months from injury or operation).
  The NRS is a modified version of the Visuel Analog Scale that consists of a segmented numerical scale with 11 points ranging from 0 to 10. The 11-point numeric scale ranges from 0 representing "no pain" to 10 representing the other pain extreme: "pain as bad as you can imagine" or "worst pain imaginable".
  This scale can be administered verbally or graphically.
Achilles tendon Total Rupture Score (ATRS) | Change from baseline to the final visit of rehabilitation (Often 6 months from injury or operation). Further assessment 12 months follow up from injury or operation.
  The Achilles tendon Total Rupture Score (ATRS) is a commonly used patient-reported outcome measure for patients with an acute Achilles tendon rupture.
  It consists of 10 questions concerning symptoms and physical activity, for which patients are asked to respond using an 11-point Likert scale (0-10). A patient scoring 0 implies major limitations/symptoms and 10 no limitations or symptoms. Answers from all 10 questions are added to a total score, with 100 being the maximum score
Thompsons test | Assessment at baseline and the final visit of rehabilitation (Often 6 months from injury or operation).
  Thompsons test (also called Simmonds squeeze test or Simmonds-Thompson test) is used in lower limb examination to test for the rupture of the Achilles tendon. The patient lies face down with feet hanging off the edge of the bed. If the test is positive, there is no movement of the foot (normally plantarflexion) on squeezing the corresponding calf, signifying likely rupture of the Achilles tendon.
Achilles Tendon Resting Angle test (ATRA) | Assessment of relative ATRA (difference between non-injured and injured leg) at baseline and the final visit of rehabilitation (Often 6 months from injury or operation). Further assessment 12 months follow up from injury or operation.
  Achilles tendon resting angle (ATRA) has been suggested and used as a surrogate measure of tendon length.
  In this test, patients are positioned in prone with the knee flexed to 90 degrees, and the passive angle that the foot falls is measured using a goniometer.
  The ATRA is the angle between the long axis of the fibula and the line from the tip of the fibula to the head of the fifth metatarsal.
  Amount of tendon elongation is defined as the difference between injured and non-injured sides (positive values indicating greater tendon length on the injured side).
Circumference of lower leg | Change from baseline to the final visit of rehabilitation (Often 6 months from injury or operation).
  Calf muscle atrophy is assessed by measuring the circumference 13 cm. below the distal apex of the patellae with a tape measure. The circumference will be recorded to the nearest 0.1 cm. and measured on both injured and the non-injured leg.
The Danish 13-item Tampa Score for Kinesiophobia (TSK-13) | Assessment at baseline and the final visit of rehabilitation (Often 6 months from injury or operation).
  The TSK is originally a 17-item self-report scale with a 4-point response scale ranging from "strongly disagree" to "strongly agree".
  Items 4, 8, 12, and 16 are reversed for scoring. A 13-item version of the scale (TSK-13) without the four reversed items has also been widely used.
  The original 17-item scale results in a total score ranging from 17 to 68 points with increasing values indicating a stronger degree of Kinesiophobia. Therefore the 13-item version results in a total score ranging from 13 to 52 points with increasing values indicating a stronger degree of Kinesiophobia.
Tegner score | Change from baseline to the final visit of rehabilitation (Often 6 months from injury or operation). Further assessment 12 months follow up from injury or operation.
  The Tegner activity score is developed as a measure of activity level. The rating system scores a person&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;s activity level between 0 and 10, where 0 is "sick leave or disability pension because of the specific problem" and 10 is "participation in competitive sports such as soccer at a national or international elite level."

OTHER OUTCOMES:
Variables that may influence on outcome: Gender | Assessment at baseline
  Assessed as female or male through the health record system
Variables that may influence on outcome: Age | Assessment at baseline
  Assessed in years through the health record system
Variables that may influence on outcome: Smoking status | Assessed at baseline
  Smoking status is described as smoking status regarding tobacco. The status is filled in by the participants with some of the patient reported outcome meassures.
  The smoking status is assessed as either smoker or non-smoker.
Variables that may influence on outcome: Body Mass Index (BMI) | Assessment at baseline
  Body weight and height are filled in by the participants with some of the patient reported outcome meassures.
  BMI is then calculated:
  Body weight in kilograms divided by the square og the height in meters.
Variables that may influence on outcome: Treatment status | Assessment after the final visit of rehabilitation (Often 6 months from injury or operation).
  Treatment status is described in either surgery or non-surgery. Assessed in through the health record system.
Variables that may influenc on outcome: Length of rehabilitation period. | Assessment after the final visit of rehabilitation (Often 6 months from injury or operation).
  Length of rehabilitation period is described in number of days through the health record system.
Variables that may influence on outcome: Number of supervised treatments in rehabilitation | Assessment after the final visit of rehabilitation (Often 6 months from injury or operation).
  Number of supervised treatments in rehabilitation is described in number of visits through the health record system.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Centre of rehabilitation Nørrebro, Copenhagen
  - Centre of rehabilitation Vanløse, Vanløse

IPD SHARING:
Plan to Share IPD: No